CLINICAL TRIAL: NCT01467791
Title: Registry of Sarcoidosis Associated Pulmonary Hypertension (RESAPH)
Acronym: RESAPH
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cincinnati (Other)
Collaborators: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Robert P Baughman, Professor of Medicine, University of Cincinnati
Other Study IDs: RESAPH 1
Record Dates: First submitted 2011-11-04; First posted 2011-11-09 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Sarcoidosis; Pulmonary Hypertension
Keywords: ambrisentan; Bosentan; Iloprost
MeSH Terms: conditions — Sarcoidosis; Hypertension, Pulmonary | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: All patients with sarcoidosis associated pulmonary hypertension
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observe patients

SUMMARY:
Registry to follow patients with sarcoidosis associated pulmonary hypertension

DETAILED DESCRIPTION:
This is a multi center registry of sarcoidosis associated pulmonary hypertension (SAPH). With this registry, the investigators will characterize the demographics, clinical course, hemodynamics, pulmonary physiology, and disease management of sarcoidosis associated pulmonary hypertension on the United States. The investigators will also compare these features to non-US sites.

ELIGIBILITY:
Inclusion Criteria:

* Patients with sarcoidosis as defined by the ATS/WASOG statement
* Patients with pulmonary hypertension as confirmed by right heart catheterization
* Patients willing to provide written informed consent

Exclusion Criteria:

* Unwillingness to provide assurance that they will complete the follow up visits for the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with sarcoidosis associated pulmonary hypertension
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-11; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Survival | 4 years
  Mortality during time of study

SECONDARY OUTCOMES:
Disease management | 4 years
  Examine initial and follow up management

CONTACTS AND LOCATIONS:
Overall Officials: Robert P Baughman, MD, Study Chair — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States